CLINICAL TRIAL: NCT02792985
Title: The Effects of Multisensory Stimulation and Enriched Environments During Post-traumatic Amnesia Following a Traumatic Brain Injury
Brief Title: Multisensory Stimulation and Enriched Environments During Post-traumatic Amnesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Guttmann (Other)
Collaborators: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014.205
Record Dates: First submitted 2016-05-08; First posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Brain Injuries, Traumatic; Confusional State; Sensory Motor System Disorder; Alteration of Cognitive Function
MeSH Terms: conditions — Brain Injuries, Traumatic; Confusion

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multisensory stimulation protocol (Experimental): The Experimental group will follow an intervention protocol.
  Interventions: Behavioral: Multisensory stimulation protocol
- Control protocol (Active Comparator): The Control group will follow the current protocol for patients in PTA at the Institut Guttmann.
  Interventions: Behavioral: Control protocol

INTERVENTIONS:
Behavioral: Multisensory stimulation protocol — Participation in occupation-based multisensory stimulation (e.g. personal care with aromatic soaps, varying water temperatures and textured sponges, drink preparation of different flavoured beverages) with a variety of different sensory stimuli (e.g. strong smells, different shapes and weights). The participant will receive two individual 30-minute therapy sessions with an Occupational Therapist.
  An enriched environment will be set up in the participant´s bedroom. It will include items that provide a range of meaningful sensory stimuli (e.g. familiar personal objects, projection of photos and known places, familiar music). The participant is encouraged to follow a timetable including regular rest breaks through out the day in their room.
  Arms: Multisensory stimulation protocol
Behavioral: Control protocol — Retraining of basic activities of daily living or participation in table top tasks and games in an individual 30 minute session or a one hour small group session with an Occupational Therapist.
  Minimal changes are made to the participant´s room (e.g. orientation board, photos of family and friends).
  Arms: Control protocol

SUMMARY:
The objective of this Phase II trial is to evaluate the feasibility of this study protocol to progress to a large-scale Phase III RCT in the future. It will also determine, with limited efficacy, the effectiveness of the multisensory stimulation intervention protocol to reduce the duration of post-traumatic amnesia (PTA), improve cognition, increase independence in activities of daily living and long term quality of life of the affected person.

Participants will be randomised into either the experimental or control group. The experimental group will follow the multisensory stimulation intervention protocol, while the control group will follow the current hospital protocol.

DETAILED DESCRIPTION:
Design: A phase II randomised controlled trial. Repeated measures of behaviour and sensory motor performance will be taken during PTA progression for all participants. The RCT involves two treatment arms and blinded assessment post-intervention at the point of PTA resolution, one month following PTA resolution, and a 6-month post-injury follow up questionnaire. The 2 treatment groups are:

1. Experimental intervention protocol: occupation-based multisensory stimulation and the use of enriched environments;
2. Control intervention protocol: standard therapy as provided by the hospital which includes re-orientation and participation in basic functional tasks.

Participants: Approximately twenty participants will be recruited from the Institut Guttmann, which is a neuro-rehabilitation hospital in Badalona, Spain.

Measures:

The evaluation tools will consist of standardised, established assessments used in brain injury rehabilitation which are detailed in the Outcome Measures section.

Procedure:

Repeated measurements of behaviour and sensory motor function corresponding to the participant's progression of PTA assessment scores will be taken. The maximum number of times a single participant will be tested during PTA is 7 times and twice again following emergence from PTA, within the first 3 days and again after 1 week. All measurements are non-invasive and provide minimal adverse risks for the participant.

Participants will be randomised into either the Experimental or Control group. Participants, their family members, and the assessor taking outcome measures at the point of PTA resolution and one-month post-resolution will be blinded to group allocation and subsequent intervention protocol. Intervention provision will occur throughout the progression of PTA with post-intervention assessment to occur within 3 days of the end of PTA, one month after coming out of PTA, and through a follow-up questionnaire to be completed by the participant and family members at 6 months post-injury. All interventions are non-invasive and do not involve any risks above those that may be incurred through participation in the standard rehabilitation process.

The Experimental group will follow an intervention protocol involving transformation of the participant´s room into a sensory stimulating enriched environment (EE) and participation in occupation-based multisensory stimulation (OBMS) during their therapy sessions with an occupational therapist. They will receive two daily 30-minute individual therapy sessions.

The control group will follow the current protocol for patients in PTA at the Institut Guttmann. This includes one 30-minute individual therapy session or one hour group therapy session with an occupational therapist and minimal changes to their room (e.g. orientation board, photos of family and friends).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of TBI
* within 6 months of their initial brain injury
* in PTA (Levels of Cognitive Function 4-6)
* appropriate visual and auditory function to observe the environment and hear instructions with or without assistive aids
* independent use of one upper limb

Exclusion Criteria:

* a previous brain injury
* illness, diseases or alcohol or drug addiction that could affect cognitive function
* having a learning disability prior to injury
* participant is out of PTA
* visual, auditory, aphasic or motor disturbance that may interfere with the ability to complete the task or participate in the sessions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-02 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Acceptability | Through study completion, up to 6 months post-injury
  The number of participants who consent to participate compared to the number who withdraw. Further understanding of this area of feasibility will be generated by family reports of satisfaction with participation in the study and reflection of the observations recorded in the project coordinator´s daily log book.
Demand | Through study completion, up to 6 months post-injury
  The percentage of eligible patients who give consent to participate in the study and the percentage that dropout after starting the study. To provide further insight of this feasibility area, analysis of demographic information of those who consent, decline or dropout will be done.
Practicality | Through study completion, up to 6 months post-injury
  Brief cost analysis to identify and measure the resources required to implement the study. A record will be taken in the project coordinator´s log book of factors observed to affect efficiency, speed, quality of implementation, or any adverse events that may occur.
Implementation | Through study completion, up to 6 months post-injury
  To measure this area of feasibility, the adherence to respective protocols for each participant will be taken including the number of days and amount of time participants attend therapy sessions. Moreover, assessment of the appropriateness of the secondary outcome measures and feasibility of the assessment protocol will be conducted.

SECONDARY OUTCOMES:
Cognitive function | Through study completion, up to 6 months post-injury
  Measured using the Neurobehavioral Cognitive Status Examination (COGNISTAT) which is a cognitive screening assessment.
Duration of PTA | Through study completion, up to 6 months post-injury
  Measured using the Westmead PTA Scale (WPTAS). PTA duration is taken to be the number of days from the date of the initial injury until the participant achieves 12/12 on the Westmead PTA Scale.
Visual perception performance | Through study completion, up to 6 months post-injury
  Measured using the Developmental Test of Visual Perception - Adolescence and Adult version to measure visual perception and visual motor integration performance.
Functional balance | Through study completion, up to 6 months post-injury
  Measured using the Berg Balance Scale.
Functional Independence | Through study completion, up to 6 months post-injury
  Measured using the Functional Independence Measure (FIM).
Level of agitation | Through study completion, up to 6 months post-injury
  Measured using the Agitated Behavior Scale (ABS).
Level of attention | Through study completion, up to 6 months post-injury
  Measured using the Moss Attention Rating Scale (MARS).

CONTACTS AND LOCATIONS:
Overall Officials: Narda Murillo, PhD, Principal Investigator — Institut Guttmann
Locations (1):
- Institut Guttmann, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No